CLINICAL TRIAL: NCT03293628
Title: Randomized Clinical Trial Comparing Two Techniques of Haemostasis After Cervical Conization With High Frequency Surgery
Brief Title: Comparing Two Techniques of Haemostasis After Cervical Conization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ricardo dos Reis, Medical Doctor, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 826/2014
Record Dates: First submitted 2017-09-04; First posted 2017-09-26 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervix Neoplasm
Keywords: cervical intraepithelial neoplasia; haemostasis; vaginal pack; Loop electrical excision procedure; randomized clinical trials; uterine cervical neoplasm
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were allocated in two arms (50 patients each): without vaginal pack (group 1 - GP1) and with vaginal pack (group 2 - GP2).Randomization was generated through a computer program creating a random entry list in the study, separating in group 1 (local application of Monsel's solution without intra-vaginal gauze buffer) and group 2 (application of Monsel's solution with intra-vaginal gauze). In this way, all patients had an equal chance of being included in both groups.
Who Masked: Participant
Masking Description: The allocation of patients to one group or another was only known moments before the surgical procedure was started.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conization With Vaginal Packing (Experimental): Experimental Arm. Haemostasis at the end of the procedure using vaginal packing and Monsel's solution.
  Interventions: Procedure: Vaginal Packing
- Conization Without Vaginal Packing (Active Comparator): Haemostasis at the end of the procedure using only Monsel's solution.
  Interventions: Procedure: Vaginal Packing

INTERVENTIONS:
Procedure: Vaginal Packing — This study will evaluate the role of vaginal packing after cervical conization as haemostasis technique

SUMMARY:
The LEEP conization is commonly used for cervical pathologies treatment. The techniques for hemostasis usually used are: cautery, Monsel's solution and vaginal pack. Actually, there is no consensus about the best technique and there is not much information that validates the use of some of that. To compare the use or not of vaginal pack as methods of hemostasis after LEEP conization for management of cervical lesions.

DETAILED DESCRIPTION:
A randomized clinical trial was conducted at Gynecology Oncology Department/Barretos Cancer Hospital for patients with indication of LEEP conization. After local IRB approval, patients were allocated in two arms (50 patients each): without vaginal pack (group 1 - GP1) and with vaginal pack (group 2 - GP2). The Monsel's solution was used in all patients. Intraoperative and postoperative outcomes will be evaluated: operative time, intraoperative and postoperative bleeding, hormonal status, age, parity and cone specimens' characteristics as well as short-term outcome were recorded and compared using Chi-square test, Fisher exact test and t-test where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Indication of cervical conization.

Exclusion Criteria:

* We excluded patients who were not treated by our department physicians or if the patient did not return for follow-up.

Ages: 19 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Vaginal bleeding until 30 days after surgery | Until 30 days after surgery
  Bleeding was assessed by the need for reintervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D Reis, MD, Principal Investigator — Hospital do Câncer de Barretos
Locations (1):
- Hospital do Câncer de Barretos, Barretos, São Paulo, Brazil